CLINICAL TRIAL: NCT02746757
Title: The Role of Glucagon Like Peptide-1 in the Protective Effect of Remote Ischemic Conditioning During Ischemia-reperfusion
Brief Title: Glucagon Like Peptide-1 in Remote Ischemic Conditioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, John Pernow, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RIPC GLP-1
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — exendin (9-39)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ischemia-reperfusion no intervention (No Intervention): Ischemia-reperfusion without intervention
- Ischemia-reperfusion with RIPC (Experimental): Ischemia-reperfusion with intervention by RIPC
  Interventions: Other: Remote conditioning
- Ischemia-reperfusion with RIPC and Ex 9-39 (Experimental): Ischemia-reperfusion with RIPC and Ex 9-39
  Interventions: Other: Remote conditioning; Drug: Exendin 9-39

INTERVENTIONS:
Other: Remote conditioning
  Arms: Ischemia-reperfusion with RIPC; Ischemia-reperfusion with RIPC and Ex 9-39
Drug: Exendin 9-39
  Arms: Ischemia-reperfusion with RIPC and Ex 9-39

SUMMARY:
The study was designed to investigate whether glucagon like peptide-1 is a mediator of protection of endothelial function induced by remote ischemic conditioning in ischemia-reperfusion

DETAILED DESCRIPTION:
The mechanism behind the cardioprotective effect of remote preconditioning is incompletely understood. Data from experimental studies suggest that a combination of humoral and neurogenic factors mediate the transition of protective signals from peripheral tissues to the myocardium. A major break-through in the understanding of the signaling was the observation that vagal nerve activation is involved. Key signaling pathways in the target organ are likely to be mediated via the vascular endothelium which is known to play an important role during the early reperfusion period. Thus, animal studies have demonstrated that RIPC stimulates endothelial nitric oxide production secondary to down-regulation of arginase. It remains unclear, however, whether RIPC via activation of endothelial nitric oxide preserves endothelial function in humans. Additional data indicate strongly that glucagon-like peptide-1 (GLP-1) provides protection against ischemia-reperfusion injury in experimental animals models as well as in clinical studies. The role of GLP-1 in the protective effect of RIPC has previously not been investigated, however. The present study was therefore designed to determine the involvement of GLP-1 in the protection induced by RIPC via endothelial activation in humans. To this end we use a model of reversible ischemia-reperfusion injury in the forearm, and the GLP-1 antagonist exendin 9-39 (Ex 9-39).

Objective To test the hypothesis that GLP-1 is a mediator of protection of endothelial function induced by RIPC in ischemia-reperfusion.

Endpoints Primary: Change in endothelium dependent vasodilatation induced by RIPC Secondary: Change in plasma GLP-1

Study subjects The study is performed on healthy volunteers 18-60 years of age. All subjects will undergo a screening including medical history and routine clinical examination, and should be free of medication. A screening blood sample includes hemoglobin, leukocyte and platelet count, fasting blood glucose, HbA1c, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides.

Methods Endothelial function is determined in the brachial artery by flow-mediated dilation (FMD). Briefly, non-invasive examination of the radial artery of the non-dominant arm is performed with a 11 MHz (output 12 MHz) linear-array transducer connected to a Vivid E9. The transducer is connected to a flexible tripod to prevent movement of the probe. Images are recorded and saved every third second at end-diastole. Baseline radial artery diameter is recorded for one minute and defined as a mean from 20 images. A blood pressure cuff is placed around the upper part of the forearm, which is inflated to 30 mmHg above systolic pressure or 200 mmHg for 5 min. The diameter of the radial artery is continuously recorded for 3 min during hyperemia following deflation of the cuff. The three frames displaying maximum dilatation at end-diastole (triggered from the ECG) are used to calculate a mean diameter. All images are analyzed with Brachial analyzer (Medical Imaging Applications, Iowa City, IA, USA). FMD is calculated as a percentage increase in diameter from baseline diameter according to the following formula: diameter following cuff deflation-baseline diameter/baseline diameter x 100. All evaluations are performed blinded. A decrease in endothelial function is an established outcome of reperfusion injury.

Study protocol After determining the basal FMD ischemia is induced by inflating a cuff to 200 mmHg on the upper arm for 20 min followed by reperfusion. FMD is determined again 20 min after the start of reperfusion . Each individual is examined on three occasions: A) ischemia-reperfusion without intervention, B) ischemia-reperfusion with intervention by RIPC, C) ischemia-reperfusion with RIPC and administration of Ex 9-39. The order of the examination is randomly assigned by drawing one of three numbers. RIPC is performed in cycles of 5 min of inflation (200 mmHg or 20 mmHg above systolic blood pressure) and 5 min deflation of an automatic blood pressure cuff around the left thigh. Two cycles are performed during ischemia and 2 cycles immediately after reperfusion. The GLP-1 receptor antagonist Ex 9-39 is administered as a bolus of 7500 pmol/kg followed by an iv infusion starting 15 min before the initial FMD and maintained until the second FMD at a rate of 500 pmol/kg/min. The dose is based on previous experiences from studies on humans.

During the experimental protocols the following blood samples are collected for analysis of glucose, insulin, GLP-1.

ELIGIBILITY:
Inclusion Criteria:

Healthy male volunteers -

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in endothelium dependent vasodilatation | 20 min post-reperfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden